CLINICAL TRIAL: NCT03215875
Title: A Randomized, Balanced, Single Dose, Two-treatment (Fed vs. Fasting), Two-period, Two-sequence, Crossover Study to Evaluate the Effects of Food on the Bioavailability of 60 mg ER Torsemide Tablet in Healthy Human Adult Subjects
Brief Title: A Food Effect Study of 60mg ER Torsemide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLCD-061-17
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Food-drug Interaction

STUDY DESIGN:
Intervention Model Description: 60mg ER Torsemide study in fed and fasting conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fed- 60mg ER Torsemide (Experimental): Adult healthy subjects will be given standardized high-fat, high-calorie meal prior to dosing
  Interventions: Drug: Fed- 60mg ER Torsemide
- Fasting- 60mg ER Torsemide (Experimental): Adult healthy subjects will fast overnight (at least 10h) prior to dosing
  Interventions: Drug: Fasting- 60mg ER Torsemide

INTERVENTIONS:
Drug: Fed- 60mg ER Torsemide — 60mg ER Torsemide will be given after high fat, high-calorie meal
  Other Names: High fat/high-calorie fed conditions
  Arms: Fed- 60mg ER Torsemide
Drug: Fasting- 60mg ER Torsemide — 60mg ER Torsemide will be given after overnight fasting
  Other Names: Fasting conditions
  Arms: Fasting- 60mg ER Torsemide

SUMMARY:
This study will evaluate the effects of a high-fat meal (food effect) on the bioavailability and pharmacokinetics of 60mg ER Torsemide tablet after single dose oral administration in healthy volunteers. The study will be conducted as a two-sequence to period crossover study to compare 60mg ER Torsemide ER bioavailability under fed and fasting conditions. 60mg ER torsemide is a new strength and dosage form.

DETAILED DESCRIPTION:
Immediate Release (IR) Torsemide is a highly effective natriuretic drug but its short duration of action is a major drawback, which allows significant post-dose sodium retention, and as consequence, limits salt loss in patients with heart failure unless dietary salt intake is severely restricted. Extended Release (ER) torsemide is being developed to address this drawback by prolonging the duration of action to increase sodium excretion even in patients who consume high salt diet. Since 60mg ER torsemide is a new strength and dosage form, this study will test 60mg ER torsemide for a food effect in healthy volunteers who are either fasting or consuming a high-fat meal (fed). The primary endpoint of the study is full pharmacokinetics measurements after a single dose of 60mg ER torsemide. The secondary endpoints are 24h sodium excretion and total urinary excretion.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female
* non-smoker
* weight ≥ 50 kg for male and ≥ 45 for female
* clinically acceptable laboratory profiles with ECG and chest x-ray performed within 6 months

Exclusion Criteria:

* participation in bioavailability/bioequivalence studies in past six months
* history of drug abuse or alcohol dependence
* history of allergies, known hypersensitivity to Torsemide and related drugs
* presence of clinically significant disorder
* suffer from high/low blood pressure (<90 and >140 mm Hg)
* positive urine drug screening, and
* history of incontinence

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Peak torsemide plasma concentration | 36 hours
  Peak plasma concentration (Cmax) (ng/ml) in fed and fasting conditions
Total torsemide plasma concentration | 36 hours
  Area under the plasma concentration versus time curve (AUC) (hr/ng/ml) in fed and fasting conditions

SECONDARY OUTCOMES:
Urinary torsemide excretion | 36 hours
  torsemide will be measured in urine over 36 hours post-dose (microgram/min)
Urinary sodium excretion | 36 hours
  36-hour sodium excretion will be measure (mmol/min)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wilcox, MD, PhD, Principal Investigator — Sarfez Pharmaceuticals, Inc.
Locations (1):
- I.E.C. Consultants, Bangalore, India

IPD SHARING:
Plan to Share IPD: No